CLINICAL TRIAL: NCT00853164
Title: A Pilot Study of Physical Activity for Improving Quality of Life in Prostate Cancer Patients on Androgen Deprivation Therapy
Brief Title: A Pilot Study of Physical Activity for Improving Quality of Life in Prostate Cancer Patients on Androgen Deprivation Therapy (ADT)
Acronym: MAP-P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 08-0318
Record Dates: First submitted 2009-02-27; First posted 2009-03-02 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; aerobic exercise; resistance training
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- aerobic exercise (Experimental): Subjects who are randomly assigned to this arm will be assigned a walking program to participate in 3 times a week for eight weeks
  Interventions: Behavioral: walking exercise
- resistence training (Experimental): Subjects who are randomly assigned to this arm will be assigned a weight training program to participate in 3 times a week for eight weeks
  Interventions: Behavioral: weight training
- Usual Care (Active Comparator): Subjects who are randomly assigned to this arm will not participate in any exercise program and will continue with usual care treatment
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: walking exercise — Subjects will be given an exercise prescription for walking 3 times a week for eight weeks
  Arms: aerobic exercise
Behavioral: weight training — participants will be given a weight training prescription to do 3 times a week for eight weeks.
  Arms: resistence training
Behavioral: Usual Care — Subjects in this arm will continue with their usual care and not start any exercise program for eight weeks.
  Arms: Usual Care

SUMMARY:
60 eligible subjects will be randomized into one of three study arms 1) aerobic exercise, 2) resistance exercise, or 3) usual care. Baseline measurements will be done on all study subjects, these measurements include: height, weight, dual energy x-ray absorptiometry (DXA) for bone mineral density and lean body mass measurements, blood will be taken to measure serum free testosterone, prostate-specific antigen (PSA), glucose, and insulin levels. Fitness will also be evaluated using a graded exercise test. Questionnaires on health and personal history will also be completed. Men randomized to the aerobic exercise treatment arm will participate in a walking program three times a week for eight weeks. The participants will start at 15 minutes per session and increase to a goal of 60 minutes per session. Men randomized to the resistance training treatment arm will participate in an eight-week program of eight strength training exercises three times per week. Men in the usual care arm will receive written materials from the American Cancer Society about coping with cancer, which includes information about participation in physical activity. At the end of the eight week intervention participants in all three study arms will complete the same questionnaires and measurements they completed at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Men with metastatic prostate cancer receiving ADT and men who have failed primary therapy and are receiving ADT.
* Men from the radiology practice who are receiving ADT as neoadjuvant therapy to primary radiotherapy (enrolled only following completion of primary radiotherapy).

Exclusion Criteria:

* Men with the following counter-indications to exercise:

  * Lower limb, bone, muscle, or joint pathology of a severity which limits their ability to be physically active.
  * A history of significant cardiac disease using criteria established by the American College of Sports Medicine ( Criteria: pain, discomfort in the chest, neck, jaw, arms, or other areas that may be due to ischemia; shortness of breath at rest or with mild exertion; ankle edema; palpitations or tachycardia; known heart murmur; unusual fatigue or shortness of breath with usual activities' syncope)
  * Other medical contraindications which would compromise participation in a lifestyle physical activity program.
  * Those who are currently physically active

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-07 (Actual); Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruiting 60 men with prostate CA on ADT to an ex intervention study w/ three arms. To determine if an ex prgm provides symptom mgt as compared to usual care,if resistance training provides symptom mgt not obtained from aerobic ex alone. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Y Wolin, ScD, Principal Investigator — Washington University School of Medicine in Saint Louis
Locations (1):
- Washington University School of medicine, St Louis, Missouri, United States